CLINICAL TRIAL: NCT04530370
Title: Efficacy and Safety of Recovered Covid 19 Plasma Transfusion to Covid 19 Severly Ill Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ossama Hamdy Salman, clinical professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ossamahamdyresearcher7
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovered covid 19 plasma (Experimental)
  Interventions: Biological: recovered covid 19 patients plasma
- controlled (Placebo Comparator)
  Interventions: Biological: recovered covid 19 patients plasma

INTERVENTIONS:
Biological: recovered covid 19 patients plasma — we transfused 150 ml of recovered covid 19 plasma to severely ill patients with confirmed covid 19 disease

SUMMARY:
The discovery of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and the outbreak of coronavirus disease 2019 (COVID-19) are causing public health emergencies. A handful pieces of literature have summarized its clinical and radiologic features, whereas therapies for COVID-19 are rather limited. To evaluate the efficacy of convalescent plasma therapy in COVID-19 patients.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a highly contagious pulmonary disease caused by a newly discovered strains of coronavirus family. The clinical pictures could range from a symptomatic to severe and can lead to hospitalization, breathing difficulties and death. Unfortunately, no vaccine or specific treatment is available so far. 1 There have been encouraging clinical researches using immunotherapy as a recent treatment modality against Covid 19 viral infections. Of particular interest, is passive immunotherapy which is the passive transfer of readymade antibodies (humoral immunity) from recovered individuals to patients in active illness. 2 Plasma of recovered patients, a classic cell transfer therapy, has been used successfully to prevent and treat many infectious diseases in the past including: H1N1 pandemic influenza A, avian influenza A (H5N1), SARS-CoV and, Ebola virus disease, MERS-CoV respiratory syncytial virus, Zika viruses, human cytomegalovirus and rabies. Unfortunately, recovered plasma did not show successful results in combating Ebola outbreak3 Neutralizing antibody from recovered SARS patients could interfere with SARS-CoV-2 from penetrating through host cells in vitro. 4 Moreover, neutralizing antibodies (NAbs) from recovered SARS-CoV patients were highly correlated, peaking at month 4 after the onset of disease, could be titrated in plasma of 90% of patients for as long as 2 years, decreasing gradually thereafter.5

SARS-CoV-2 is a member of β-coronavirus family. It is a single-stranded RNA genome consists of 30 kb nucleotides, which transcript 4 main structural proteins: spike (S), membrane (M), envelope (E), and nucleocapsid (N) proteins. The virus characteristic appearance stems from, the S protein which is club shape glycoprotein radiating in a crown like configuration. 6 Genome researches have shown that interlocking between the receptor-binding domain of S protein and the angiotensin-converting enzyme 2 (ACE2) facilitates SARS-CoV-2 entry into the host cells. 7 The similarity of the receptor-binding sites between SARS-CoV-2 and SARS-CoV explains their shared pathogenicity and biological traits. Moreover, both covid-19 and SARS share common clinical (fever, cough, body aches, and dyspnea) and typical radiological manifestations (multifocal ground-glass opacities (GGOs) and subsegmental areas of consolidation). 8 Nevertheless, both viruses are highly contagious with incubation period range from several days to two weeks.

Patients with SARS-CoV-2 infection produce different antibodies against different viral antigenic proteins (epitomes), and some of these antibodies mediate their action by virus neutralization or by phagocytosis and antibody gated cell toxicity.9 There have been published studies claiming successful patient outcome after transfusion of recovered plasma. One study showed improved clinical pictures, higher discharge rate. 10 Another study demonstrated that viral RNA disappeared in patient serums a week post transfusion. 11 Another study compared the clinical improvement of recovered plasma transfusion with steroids in SARS patients with critical condition. They observed that recovered plasma patients had a high hospital discharge rate, better clinical outcome than the steroid group, with no transfusion related unwanted effects.12 A large meta-analysis of 1703 influenza pneumonia patients who had been transfused recovered plasma, showed a marked decrease of viral load and 21% decrease in mortality. 13 There are fast growing numbers of new COVID-19 cases every day, and disease-related morbidity and mortality is increasing. The purpose of our study was to test the efficacy and safety of transfusing plasma from patients who have recovered from COVID-19, to patients with COVID-19 in severe condition.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years, with confirmed laboratory covid-19, and have one or more of the following 4 conditions:

  * 1. respiratory frequency ≥ 30/min,
  * 2. blood oxygen saturation ≤ 93% on room air,
  * 3. partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300 mmHg,
  * 4. pulmonary infiltrates occupying more than 50% of both lungs.

Exclusion criteria

* Any patient with prior allergic history to plasma or
* allergy to plasma products or
* septic shock or
* multiple organ failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Satisfactory outcome | 5 days
  Patients' response to recovered Covid 19 plasma (RCP) during 5 days after transfusion, was our primary goal. It was categorized into either satisfactory or unsatisfactory outcomes. We defined satisfactory outcome as two or more of the following 4 conditions/ or otherwise unsatisfactory: 1. respiratory frequency < 30/min, 2. Sustain blood oxygen saturation ≥93% on room air, 3. partial pressure of arterial oxygen to fraction of inspired oxygen ratio > 300 mmHg, 4. Regression of pulmonary infiltrates occupying less than 50% of both lungs.

CONTACTS AND LOCATIONS:
Overall Officials: Gad s Gad, MD, Study Chair — South Valley University
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969